CLINICAL TRIAL: NCT04722601
Title: A Multicenter, Single-Arm, Phase I/II Dose Finding and Efficacy Study of Venetoclax, CC-486, and Obinutuzumab in Minimally-Pretreated Follicular Lymphoma
Brief Title: A Dose-Finding and Efficacy Study of Venetoclax, CC-486, and Obinutuzumab in Follicular Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-0986
Record Dates: First submitted 2020-11-02; First posted 2021-01-25 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma, FL
MeSH Terms: conditions — Lymphoma, Follicular | interventions — venetoclax; obinutuzumab; cc-486; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose (Experimental): Phase 1/the dose-finding arm of this study will use three dose levels (a starting dose, second dose and highest dose) of the venetoclax, CC-486 and obinutuzumab regimen. If participants in group 1 don't experience severe negative side effects to the starting dose of the regimen, then more participants will be assigned to groups 2 and 3 to take higher doses until the safest/ most tolerable dose is found.
  Group 1/ Dose Level 1:
  Participants in group 1 will receive a three-drug regimen of venetoclax, CC-486, and obinutuzumab at a starting dose used in previous human studies. Participants in this group will receive:
  * Venetoclax:
    400 mg on days 1-28
  * CC-486:
    200 mg on days 1-14
  * Obinutuzumab:
    1000 mg on days 1, 8 and 15 of cycle 1, and on day 1 of each following cycle.
  Treatment using these three study drugs (venetoclax, CC-486, and obinutuzumab) will be given in 12 consecutive cycles that run for 28 days during each cycle (336 days).
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab; Drug: CC-486
- Phase 2 (Efficacy Arm/ Expansion Cohort) (Experimental): Participants in this arm will help test the efficacy of the three-drug regimen and dose established in the phase 1 of the study. Participants will take two drugs (venetoclax and CC-48) used in the same three-drug regimen during the first phase of this study. These two drugs will be paired together by themselves and given to participants in the expansion cohort before obinutuzumab (a third drug) is added during cycle 4 of treatment.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab; Drug: CC-486
- Phase 1(Dose-Finding Arm): Group 2 - Dose Level 2 /Second Dose (Experimental): Participants in group 2 will receive a three-drug regimen of venetoclax, CC-486, and obinutuzumab at the second highest dose (dose level 2) set by doctors leading the study. Participants in this group will receive:
  * Venetoclax:
    600 mg on days 1-28
  * CC-486:
    200 mg on days 1-14
  * Obinutuzumab:
    1000 mg on days 1, 8 and 15 of cycle 1, and on day 1 of each following cycle.
  Treatment using these three study drugs (venetoclax, CC-486, and obinutuzumab) will be given in 12 consecutive cycles that run for 28 days during each cycle (336 days).
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab; Drug: CC-486
- Phase 1 (Dose-Finding Arm) - Group 3 - Dose Level 3/ Highest Dose (Experimental): Participants in group 3 will receive a three-drug regimen of venetoclax, CC-486, and obinutuzumab at the highest dose (dose level 3) set by doctors leading the study. Participants in this group will receive:
  * Venetoclax:
    800 mg on days 1-28
  * CC-486:
    200 mg on days 1-14
  * Obinutuzumab:
    1000 mg on days 1, 8 and 15 of cycle 1, and on day 1 of each following cycle.
  Treatment using these three study drugs (venetoclax, CC-486, and obinutuzumab) will be given in 12 consecutive cycles that run for 28 days during each cycle (336 days).
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab; Drug: CC-486
- Phase 1 (Dose-Finding Arm) - Group 4 - Lower Dose Level 1 (Experimental): Participants in this group will received a lower dose of the three-drug regimen using venetoclax, CC-486 and obinutuzumab set by doctors leading the study. Inclusion in this group is optional and based on whether the participant reports serious adverse events/side effects in response to a higher dose of the regimen. If participants are included in this group, they will receive:
  * Venetoclax:
    400 mg on days 1-28
  * CC-486:
    150 mg on days 1-14
  * Obinutuzumab:
    1000 mg on days 1, 8 and 15 of cycle 1, and on day 1 of each following cycle.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab; Drug: CC-486
- Phase 1 (Dose-Finding Arm) - Group 5 - Lower Dose Level 2 (Experimental): Participants in this group will received the second lowest dose of the three-drug regimen using venetoclax, CC-486 and obinutuzumab set by doctors leading the study. Inclusion in this group is optional and based on whether the participant reports serious adverse events/side effects in response to a higher dose of the regimen. If participants are included in this group, they will receive:
  * Venetoclax:
    400 mg on days 1-10 only
  * CC-486:
    150 mg on days 1-14
  * Obinutuzumab:
    1000 mg on days 1, 8 and 15 of cycle 1, and on day 1 of each following cycle.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab; Drug: CC-486

INTERVENTIONS:
Drug: Venetoclax — A drug used with other drugs to treat acute myeloid leukemia that is newly diagnosed. It is used in adults who are 75 years and older or in adults who cannot be treated with other anticancer drugs. Venetoclax is also used to treat chronic lymphocytic leukemia and small lymphocytic lymphoma in adults. It is also being studied in the treatment of other types of cancer.
  Other Names: Venclexta; Venclyxto
Drug: Obinutuzumab — Obinutuzumab is a prescription medicine that can be used in combination with other cancer medicines to treat follicular lymphoma (a type of non-Hodgkin lymphoma), or to help delay the progression of this disease.
  Other Names: Gazyva
Drug: CC-486 — An oral form of azacitidine (a standard chemotherapy drug).
  Other Names: azacitidine

SUMMARY:
This study focuses on finding a safe and tolerable dose for a three-drug regimen that combines venetoclax (Venclexta Ⓡ), CC-486 (also known as oral azacitidine) and obinutuzumab (Gazyva Ⓡ) to treat cancer participants who have minimally pretreated follicular lymphoma and have experienced disease progression despite trying previous cancer therapies. If a safe and tolerable drug dose can be found in the first phase of the study, doctors leading the study will launch a second phase of the study within an expansion cohort. Participants in this expansion cohort will receive the dose established in the first phase of the study to determine the efficacy of the regimen/ established dose. Participants in the expansion cohort will also receive the same study drugs from the first phase of the study, but in a different order/combination (first pairing the two oral drugs, CC-486 and venetoclax, then adding the third drug, obinutuzumab to treatment). The end goal of this research is to establish a new chemotherapy-sparing treatment option for patients with follicular lymphoma that is just as effective (or better) than current standard of care options.

ELIGIBILITY:
INCLUSION CRITERIA

Participants are eligible to be included in the study if all of the following criteria apply:

1. Male and female participants who are at least 18 years old with a medically confirmed diagnosis of grade 1-3a follicular lymphoma by 2017 World Health Organization criteria. A prior tissue or bone marrow biopsy may be used to confirm diagnosis if collected within 90 days of initiating therapy.
2. Treatment-naive (you have never had treatment for your cancer) or if you have received treatment, you have received fewer than two prior lines of anti-CD20 monotherapy consisting of a total of 16 or fewer doses.
3. Must have Stage II-IV disease on screening PET imaging with measurable disease, according to Lugano Classification. Measurable disease will be defined as at least one lesion that can be accurately measured in at least two dimensions and quantifiable avidity ( a tumor containing antibodies that have a higher rate/stability of binding with an antigen) to F-fluorodeoxyglucose (also known as "FDG" - a glucose analogue that can be high in cancerous tumors) . Minimum measurement must be >15 mm in the longest diameter by >10 mm in the short axis.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less as defined in Appendix B. Performance status must be evaluated within 28 days prior to treatment initiation.
5. There must be a clear way to indicate that you need treatment, either by meeting one or more of the Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria for treatment (Brice et al. 1997), the existence of cancer-related pain or other uncontrollable symptoms. Study participant whose need for treatment can be supported by the judgment of a primary oncologist based on the pace of their disease progression/other clinical criteria are also eligible for the study. Study participants must have documented progression of disease.
6. Not be a candidate for standard-of-care chemoimmunotherapy in the judgment of the primary oncologist OR standard chemoimmunotherapy was discussed with the primary oncologist and declined by the participant.
7. A male participant must agree to use contraception during the treatment period of this study, and for at least 90 days after the last dose of venetoclax or 18 months after the last dose of obinutuzumab, whichever is longer, and refrain from donating sperm during this period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of obinutuzumab to avoid exposing the embryo.
8. A female participant is eligible to participate if she is not pregnant, breastfeeding, and at least one of the following conditions applies:

   * She is not a woman of childbearing potential
   * She is a woman of childbearing potential who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of venetoclax or 18 months after the last dose of obinutuzumab, whichever is longer.
   * Participants must have a negative pregnancy test within 72 hours of beginning treatment if they are women of childbearing potential.
9. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
10. Have adequate organ function that can be confirmed by clinical laboratory values within 28 days prior to treatment initiation.

EXCLUSION CRITERIA

Participants are excluded from the study if any of the following criteria apply:

1. A a woman of childbearing potential who has a positive urine pregnancy test within 72 hours prior to treatment allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for the subject to start receiving study medication.
2. Has received any prior systemic therapy other than anti-CD20 monoclonal antibody or radiotherapy prior to the first dose of study medication. Subjects must not have had a prior dose of anti-CD20 monoclonal antibody therapy within 28 days prior to the first dose of study medication.
3. Known hypersensitivity or allergy to any of the study drugs, xanthine oxidase inhibitors and/or rasburicase, mannitol, murine products, or any components of the drug formulations.
4. History of severe allergic or anaphylactic reaction to humanized or murine monoclonal antibodies.
5. History of other malignancy that could affect compliance with the study or interpretation of results such as:

   * Participants with a history of basal or squamous cell carcinoma or stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible.
   * Participants with a malignancy that has been treated with surgery alone with the intent to cure the participant will also be excluded. Individuals in documented remission without treatment for 2 years prior to enrollment may be included at the discretion of the doctor leading the study.
6. Has medical/clinical evidence of transformation to an aggressive lymphoma subtype including grade 3b Follicular Lymphoma.
7. Has received the following agents within 7 days prior to the first dose of venetoclax:

   * Steroid therapy for anti-neoplastic intent
   * A strong or moderate Cytochrome P450 3A (abbreviated as "CYP3A" inhibitor).
   * CYP3A inducers
   * Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of venetoclax
   * P-glycoprotein (P-gp) inhibitors or narrow therapeutic index P-gp substrates
8. Evidence of significant, uncontrolled diseases that could affect the participant's ability to fulfill their role in the study/ protocol or interpretation of results or that could increase risk to the participant, including renal disease that would preclude chemotherapy administration or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).
9. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1. Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment) will result in study exclusion. Caution should be exercised when considering the use of any of the study medication in participants with a history of recurring or chronic infections.
10. Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
11. Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody. Participants who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation. Participants with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These participants must be willing to undergo monthly HBV DNA testing.
12. Receipt of live-virus vaccines within 30 days prior to the initiation of study treatment
13. Malabsorption syndrome, inability to swallow a large number of pills, or other condition that precludes enteral route of administration.
14. A history of progressive multifocal leukoencephalopathy (PML) or known prior infection with the John Cunningham (JC) virus.
15. Significant active cardiac disease within the previous 6 months including New York Heart Association class 4 heart failure, unstable angina, or myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated. Only 2 participants were enrolled at the starting dose.
Period: Overall Study
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase I Objective: Maximum Tolerated Dose of Venetoclax and CC-486 As Assessed by Rate of Reported Dose Limiting Toxicities (Side Effects) According to CTCAE Criteria Version 5
Description: The maximum tolerated dose of venetoclax and CC-486 in patients with minimally pre-treated follicular lymphoma. Doctors leading the study will find the maximum tolerated dose by assessing the rate of serious side effects (known as "dose limiting toxicities") according to the NCI Common Terminology Criteria (CTCAE) for Adverse Events Version 5.
Time Frame: 336 days (the duration of phase 1 treatment)
Population: Data not collected
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 0

2. Primary Outcome: Phase I Objective: Number of Participants Who Discontinue Venetoclax, CC-486 and Obinutuzumab Regimen Due to Reported Side Effects as Assessed by CTCAE Criteria Version 5
Description: The number of participants who discontinue the three-drug regimen of venetoclax, CC-486, and obinutuzumab during phase 1 of the study due to serious side effects (grade 3/4) as assessed by the NCI Common Terminology Criteria (CTCAE) for Adverse Events Version 5.
Time Frame: 336 days (duration of phase 1 treatment)
Population: Data not collected
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 0

3. Primary Outcome: Phase I Objective: Number of Participants Taking Venetoclax, CC-486 and Obinutuzumab Who Report Serious Side Effects As Assessed by CTCAE Version 5
Description: The number of participants who report serious side effects in response to the three-drug regimen of venetoclax, CC-486 and obinutuzumab during phase 1 treatment. Serious side effects will be defined as grade 3/ 4 according to criteria set by the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.
Time Frame: 336 days (duration of phase 1 treatment)].
Population: Data not collected
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 0

4. Primary Outcome: 4. Phase II Objective: Number of Participants Who Do Not Show Signs of Cancer After Taking CC-486 and Obinutuzumab (Oral Therapies) As Assessed by PET/CT Whole Body Scan (Based on Lugano Criteria)
Description: The number of participants who do not show detectable signs of cancer (also known as "complete response") after taking combined CC-486 and obinutuzumab as assessed by positron emission tomography (PET scan) based on Lugano criteria.
Time Frame: 336 days (duration of phase 1 treatment)
Population: Data not collected
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase II Objective: The Length of Time That Half of Participants in the Expansion Group Are Alive After Receiving Phase 1 Dose of Treatment As Assessed at End of Study and 5 Years After Study is Complete
Description: The length of time that half of the participants in the expansion/phase II study group are alive after taking the maximum tolerated dose established in the first phase of the study. This time, also known as "median overall survival," will be documented at the end of the study and five years after study completion.
Time Frame: 55 months (at study conclusion) and 5 years after end of study
Population: Data not collected
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase II Objective: The Average Length of Time Participants Treated at Phase 1 Dose Live With Follicular Lymphoma Without Symptoms of Cancer Worsening As Assessed at End of Study and 5 Years After Study is Complete
Description: The average length of time study participants in the expansion/phase II group of the study live with follicular lymphoma, but it does not get worse (also known as "median progression-free survival" of participants). This time will be assessed at the conclusion of study and five years after study completion.
Time Frame: 55 months (at study conclusion) and 5 years after end of study
Population: Data not collected
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase II Objective: Number of Participants Who Do Not Show Signs of Follicular Lymphoma After Venetoclax and CC-486 As Assessed by PET Scan (Based on Lugano Criteria)
Description: Number of participants in phase II group who do not show signs of follicular lymphoma after receiving three cycles of venetoclax + CC-486 (combined oral therapy). This will be assessed by positron emission tomography (PET scan) based on Lugano criteria.
Time Frame: 84 days (three cycles of combined oral therapies venetoclax and CC-486 oral
Population: Data not collected
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase II Objective: Number of Participants Who Do Not Show Signs of Follicular Lymphoma 30 Months After Treatment As Assessed by PET Scan (Based on Lugano Criteria
Description: Number of participants who do not show signs of follicular lymphoma (also known as "complete response rate") 30 months after starting treatment. This will be assessed by positron emission tomography (PET scan) based on Lugano criteria.
Time Frame: 30 months and 336 days (treatment period); approximately 3.4 years
Population: Data not collected
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose (N=2)
Neutrophil count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1(Dose-Finding Arm): Group 1 - Dose Level 1 / Starting Dose (N=2)
Alkaline phosphatase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT04722601/Prot_SAP_000.pdf